CLINICAL TRIAL: NCT03428516
Title: Decrease in Sympathetic Tone in OSA Patients: Is CPAP More Effective Than APAP ?
Brief Title: Decrease Obstructive Sleep Apnea (OSA) Sympathetic Tone : Impact of APAP vs CPAP
Acronym: APAP-CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); ResMed (Industry); Agir pour les maladies chroniques (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2017-A02937-46
Record Dates: First submitted 2018-01-17; First posted 2018-02-09 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2022-07

CONDITIONS: Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed CPAP (Experimental): CPAP always deliver air with the same pressure
  Interventions: Device: Fixed CPAP
- Auto-adjusting CPAP (Active Comparator): Auto-CPAP changes the pressure delivered depending on events detected at any time (apnea, hypopnea …) and applies the lowest pressure required to eliminate events.
  Interventions: Device: Auto-adjusting CPAP

INTERVENTIONS:
Device: Fixed CPAP — CPAP is a device that applies continous fixed positive pressure to the airways in order to keep them opened during sleep
  Arms: Fixed CPAP
Device: Auto-adjusting CPAP — Auto-adjusting CPAP is a device that applies auto-adjusting continous positive pressure to the airways in order to keep them opened during sleep
  Arms: Auto-adjusting CPAP

SUMMARY:
The present study aims to compare muscle sympathetic neural activity by microneurography after one month treatment of fixed versus auto-adjusting CPAP treatment and its impact on arterial blood pressure

DETAILED DESCRIPTION:
Background: Sleep apnea syndrome (SAS) currently affects 10% of general population. It is characterized by the occurrence during the sleep of the upper airways closure which cause repeated asphyxia. It is a public health problem due to its cardiometabolic complications. Indeed, the absence of SAS treatment increases cardiovascular mortality by 12% at 10 years.

The main physiopathological mechanism is the activation of cardiovascular sympathetic control (the short-term regulation of blood pressure which bring in the sympathetic nervous system) An exposure to intermittent chronic hypoxia (caused by SAS) bring an increased of muscle sympathetic nerve activity (MSNA) contributing to elevated blood pressure Continuous Positive Airway Pressure (CPAP) can partly reduce this risk by decreasing elevation of blood pressure caused by the SAS. It has recently been demonstrated that all CPAP devices are not equivalent. Indeed, the auto-adjusted CPAP treatment induces a reduction in blood pressure lower than the reference treatment fixed CPAP.

To this extent it is interesting to conduct a new randomized trial comparing these two treatments with vascular sympathetic tone. This will be assessed by peroneal microneurography recording.

Objective: Compare Muscle Sympathetic Neural Activity (MSNA) by microneurography after one month of fixed versus auto-adjusted CPAP treatment in OSA patients naive from pressure therapy Methods: Prospective study, single-site, randomized, double-blind, parallel, one month controlled trial. After the diagnosis of sleep apnea, patients will be randomized for one month treatment with fixed ou auto-adjusting CPAP. Measurements of MSNA, heart rate variability and catecholamines will be held before and after treatment.

An interim analysis will be performed after the inclusion of 24 patients based on group sequential design.

Assuming an α error of 5%, a statistical power of 80%, and a unilateral situation : 34 patients per arm will be needed to be enrolled in the study. The enrollment target for the study will be reviewed and may be refined following the study interim analysis and taking account 20% of study drop-out.

ELIGIBILITY:
Inclusion Criteria:

* patient with OSA (AHI ≥20 / h)
* patient with daytime sleepiness
* naive of any pressure treatment of OSA
* patient able to provide written informed consent
* not a vulnerable person or legally protected adult.

Exclusion Criteria:

* pregnancy
* Person deprived of liberty or subject to a legal protection measure.
* Patient with serious heart failure (According to investigator judgment)
* patient with central sleep apnea index above 20% of AHI
* Patient with a significant intercurrent pathology that can influence the results. (According to investigator judgment).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Sympathetic tone (MSNA) | Change from baseline after one month of intervention
  Change from Baseline Sympathetic tone at 1 months

SECONDARY OUTCOMES:
24 hours Systolic Blood pressure (AMBP) | Change from baseline after one month of intervention
  Change from Baseline in 24 hours ambulatory systolic blood pressure
Systolic Blood pressure (office) | Change from baseline after one month of intervention
  Clinical BP on 3 occasions, SBP and BP will be assessed. Mean BP calculated as DBP+1/3(SBP-DBP)
Diastolic Blood pressure (office) change after 1 month | Change from baseline after one month of intervention
  Clinical BP on 3 occasions, SBP and BP will be assessed. Mean BP calculated as DBP+1/3(SBP-DBP)
Mean Blood pressure (office) | Change from baseline after one month of intervention
  Clinical BP on 3 occasions, SBP and BP will be assessed. Mean BP calculated as DBP+1/3(SBP-DBP)
Catecholamines (epinephrine) | Change from baseline after one month of intervention
  24h urine samples will be collected and acidified with acetic acid, stored at -20°C until analysis. Catecholamines (epinephrine, norepinephrine, and dopamine) will be measured in one milliliter of urine by high-performance liquid chromatography with electrochemical detection (CoulArray® Detector from ESA- Dionex, Chelmsford, USA).
Norepinephrine) | Change from baseline after one month of intervention
  24h urine samples will be collected and acidified with acetic acid, stored at -20°C until analysis. Catecholamines (epinephrine, norepinephrine, and dopamine) will be measured in one milliliter of urine by high-performance liquid chromatography with electrochemical detection (CoulArray® Detector from ESA- Dionex, Chelmsford, USA).
Dopamine (Catecholamine) | Change from baseline after one month of intervention
  24h urine samples will be collected and acidified with acetic acid, stored at -20°C until analysis. Catecholamines (epinephrine, norepinephrine, and dopamine) will be measured in one milliliter of urine by high-performance liquid chromatography with electrochemical detection (CoulArray® Detector from ESA- Dionex, Chelmsford, USA).
High-frequency component of Heart rate variability | Change from baseline after one month of intervention
  We will use these mathematical methods to analyze a signal over time: temporal analysis, Fourier transformation and wavelet transformation.
  High-frequency (HF) translates fluctuations in parasympathetic activity to cardiac destination, modulated by ventilatory characteristics (frequency, courant volume).
Low frequency component of Heart rate variability | Change from baseline after one month of intervention
  We will use these mathematical methods to analyze a signal over time: temporal analysis, Fourier transformation and wavelet transformation.
  Low frequency (LF) is classically considered to reflect the activity of the sympathetic system rather than the parasympathetic system.
24 hours Diastolic blood pressure change (AMBP) | Change from baseline after one month of intervention
  ambulatory measurements over 24h
24 hours Mean Blood pressure (AMBP) | Change from baseline after one month of intervention
  ambulatory measurements over 24h

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Tamisier, MD, PhD, Principal Investigator — University Grenoble Alps
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pepin JL, Tamisier R, Baguet JP, Lepaulle B, Arbib F, Arnol N, Timsit JF, Levy P. Fixed-pressure CPAP versus auto-adjusting CPAP: comparison of efficacy on blood pressure in obstructive sleep apnoea, a randomised clinical trial. Thorax. 2016 Aug;71(8):726-33. doi: 10.1136/thoraxjnl-2015-207700. Epub 2016 Apr 18. PMID 27091542
- [Derived] Treptow E, Pepin JL, Bailly S, Levy P, Bosc C, Destors M, Woehrle H, Tamisier R. Reduction in sympathetic tone in patients with obstructive sleep apnoea: is fixed CPAP more effective than APAP? A randomised, parallel trial protocol. BMJ Open. 2019 Apr 4;9(4):e024253. doi: 10.1136/bmjopen-2018-024253. PMID 30948567